CLINICAL TRIAL: NCT01681173
Title: Investigation of the Effect of Insoluble Dietary Fiber on Carbohydrate and Lipid Metabolism and the Prevention of Diabetes Mellitus Type 2 in Subjects With Impaired Glucose Tolerance
Brief Title: OPTIFIT-Optimal Fiber Trial for Diabetes Prevention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: German Institute of Human Nutrition (Other)
Collaborators: Charite University, Berlin, Germany (Other); German Diabetes Foundation, Munich, Germany (Unknown); Ernst von Bergmann Hospital (Other); University Hospital Tuebingen (Other)
Responsible Party: Principal Investigator, Prof. Dr. med. Andreas F. H. Pfeiffer, Chief, Department of Clinical Nutrition, German Institute of Human Nutrition
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: DDS-FKZ 232/11/08
Record Dates: First submitted 2012-09-05; First posted 2012-09-07 (Estimated); Last update posted 2015-02-05 (Estimated); Status verified 2015-02

CONDITIONS: Diabetes; Nutrition Disorders; Obesity; Overweight; Metabolic Syndrome x; Body Weight; Glucose Metabolism Disorders; Metabolic Diseases
Keywords: Nutritional support; Diet therapy; Diabetes prevention; Insoluble fiber; Healthy life style; Weight loss
MeSH Terms: conditions — Diabetes Mellitus; Nutrition Disorders; Obesity; Overweight; Metabolic Syndrome; Body Weight; Glucose Metabolism Disorders; Metabolic Diseases; Weight Loss | interventions — Dietary Fiber

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Drink enriched in fibers (Experimental): 7,5g enriched fiber drinks, BID
  Interventions: Dietary Supplement: Fiber
- Placebo drink (Experimental): Placebo drink, BID
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Fiber — 200ml drinks enriched with 7,5g of fiber (90% insoluble fiber, 10% soluble fiber), BID, over 24 months
  Arms: Drink enriched in fibers
Dietary Supplement: Placebo — 200ml Placebo, BID, over 24 months
  Arms: Placebo drink

SUMMARY:
High intake of insoluble fiber is strongly associated with a reduced incidence of diabetes and cardiovascular events in prospective observation studies. Our primary objective is to compare a life style diabetes prevention program(PRAEDIAS) with and without added insoluble fibers in its effectiveness to prevent incident diabetes type 2 in high risk individuals with impaired glucose tolerance. Subjects with IGT not willing to participate in the intervention will be used as independent controls. Secondary aims are to identify mechanisms of action with regard to body composition, anti-inflammatory and metabolic effects of fibers. We propose a randomized, prospective intervention study. The results will be of general relevance for guidance of fiber intake in the population and will help the food industry to design healthy high fiber foods. Fiber can be added at low cost to numerous foods. Increased fiber intake may therefore provide a simple non-cognitive prevention strategy effective at the population level.

DETAILED DESCRIPTION:
The overall objective is to investigate whether insoluble fibers added to standard nutrition can reduce the progression of impairment of glucose metabolism in a high risk population with impaired glucose metabolism. Large prospective cohort studies clearly show that mainly insoluble cereal fiber from whole grains is associated with reduced risk of type 2 diabetes and cardiovascular disease. However, there is a lack of evidence from prospective intervention studies targeted to evaluate the potential of dietary fibers to reduce diabetes and cardiovascular disease as recently stated by the Cochrane Foundation. Dietary fiber intake is generally much lower than currently recommended, which may in part be related to side effects of whole grain nutrients and their gustatory properties. Intestinally uncomfortable effects are at least partly related to fermentation which is much less induced by insoluble non-fermentable fibers than by soluble fermentable fibers. The prospective demonstration of beneficial effects of insoluble fibers in preventing diabetes type 2 will allow detailed nutritional recommendations. This may serve to support the consumption of metabolically beneficial constituents of fiber-rich diets and help to increase fiber intake by high fiber natural nutrients or everyday nutrients enriched in insoluble natural fibers.

ELIGIBILITY:
Inclusion Criteria:

* Impaired glucose tolerance
* Age>18years old
* both gender

Exclusion Criteria:

* Diabetes type 1 and type 2
* chronic or malignant disease
* Intake of metabolic influence drugs
* Food allergies, fiber intolerance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2010-05; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Change of 2h-postprandial blood glucose from IGT to diabetes mellitus type 2 or normal glucose tolerance (NGT) | 0, 12, 24 months
  Change of the glucose metabolism (OGTT)

SECONDARY OUTCOMES:
Change of insulin sensitivity | 0, 12, 24 months
  Measurement by HOMA and OGIS from the OGTT
Change of insulin secretion | 0, 12, 24 months
  Measurement by the OGTT
Expression of inflammatory markers in blood | 0, 6, 12, 18, 24 months
  CRP, leukocytes, adipocytokines
Biometric data | 0, 6, 12, 18, 24 months
  Nutritional impact of blood pressure, anthropometry (body weight and body composition)
Assessment of cognitive performance | 0, 12, 24 months
Development of indices for the prediction of fat mass | 0, 12, 24 months
  Change of fat fraction in liver, abdominal and in the total body fat measuring by MRI/H1-spectroscopy
Determination of gene expression in adipose tissue | 0, 12, 24 month
  Determination of inflammatory and other transcripts in sc adipose tissue in a fat biopsy.

CONTACTS AND LOCATIONS:
Overall Officials: Andreas FH Pfeiffer, Prof., Principal Investigator — German Institute of Human Nutrition Potsdam-Rehbruecke
Locations (2):
- Germany (2):
  - German Instiute of Human Nutrition, Potsdam-Rehbruecke, Nuthetal
  - Charite University, Berlin, State of Berlin

REFERENCES:
- [Derived] Kabisch S, Montagna F, Honsek C, Kemper M, Gerbracht C, Arafat AM, Birkenfeld AL, Dambeck U, Osterhoff MA, Weickert MO, Floel A, Pfeiffer AFH. Effects of lifestyle intervention and supplementation with insoluble oat fiber on cognitive functions in patients with prediabetes: a secondary analysis of the Optimal Fiber Trial. Front Nutr. 2026 Jan 16;12:1699958. doi: 10.3389/fnut.2025.1699958. eCollection 2025. PMID 41624204
- [Derived] Honsek C, Kabisch S, Kemper M, Gerbracht C, Arafat AM, Birkenfeld AL, Dambeck U, Osterhoff MA, Weickert MO, Pfeiffer AFH. Fibre supplementation for the prevention of type 2 diabetes and improvement of glucose metabolism: the randomised controlled Optimal Fibre Trial (OptiFiT). Diabetologia. 2018 Jun;61(6):1295-1305. doi: 10.1007/s00125-018-4582-6. Epub 2018 Feb 28. PMID 29492637